CLINICAL TRIAL: NCT07100106
Title: A Phase Ib/II Multicenter, Open-Label, Randomized Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-4198 Alone and in Combination With Giredestrant in Comparison With Abemaciclib and Giredestrant in Participants With Locally Advanced or Metastatic Estrogen Receptor-Positive, HER2-Negative Breast Cancer Who Have Previously Progressed During or After a CDK4/6 Inhibitor
Brief Title: A Study to Evaluate the Effect of GDC-4198 Alone and in Combination With Giredestrant Versus Abemaciclib and Giredestrant in Participants With Locally Advanced or Metastatic Estrogen Receptor-Positive (ER+), Human Epidermal Growth Factor Receptor-Negative (HER2-) Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche (China) Holding Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO46021; 2025-521128-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-31; First posted 2025-08-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase Ib: Dose-Finding Stage (Experimental): Participants will receive GDC-4198 as monotherapy and in combination with giredestrant, 30 milligrams (mg), orally, daily, as per a pre-defined dosing regimen during each cycle until unacceptable toxicity or disease progression and/or loss of clinical benefit. (1 cycle=28 days).
  Interventions: Drug: GDC-4198; Drug: Giredestrant
- Phase II: Arm A (Experimental): Participants will receive GDC-4198, higher dose, in combination with giredestrant, 30 mg, orally, daily, as per a pre-defined dosing regimen during each cycle until unacceptable toxicity or disease progression and/or loss of clinical benefit. (1 cycle=28 days).
  Interventions: Drug: GDC-4198; Drug: Giredestrant
- Phase II: Arm B (Experimental): Participants will receive GDC-4198, lower dose, in combination with giredestrant, 30 mg, orally, daily, as per a pre-defined dosing regimen during each cycle until unacceptable toxicity or disease progression and/or loss of clinical benefit. (1 cycle=28 days).
  Interventions: Drug: GDC-4198; Drug: Giredestrant
- Phase II: Arm C (Experimental): Participants will receive abemaciclib, 150 mg twice daily, in combination with giredestrant, 30 mg, orally, daily, as per a pre-defined dosing regimen during each cycle until unacceptable toxicity or disease progression and/or loss of clinical benefit. (1 cycle=28 days).
  Interventions: Drug: Giredestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: GDC-4198 — GDC-4198 will be administered orally.
  Other Names: RGT-419B; RO7840734
  Arms: Phase II: Arm A; Phase II: Arm B; Phase Ib: Dose-Finding Stage
Drug: Giredestrant — Giredestrant will be administered orally.
  Other Names: GDC-9545; RO7197597
Drug: Abemaciclib — Abemaciclib will be administered orally.
  Arms: Phase II: Arm C

SUMMARY:
The purpose of this study is to assess the safety of GDC-4198 alone and in combination with giredestrant and also the efficacy of GDC-4198 + giredestrant versus abemaciclib + giredestrant in participants with locally advanced or metastatic ER+, HER2- breast cancer. The study consists of 2 phases: Phase Ib and Phase II. Phase Ib will evaluate the safety and pharmacokinetics (PK) of GDC-4198 alone and in combination with giredestrant. Phase II stage will compare the activity and safety of GDC-4198 and giredestrant with abemaciclib and giredestrant.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed adenocarcinoma of the breast that is locally advanced or metastatic.
* Previously documented ER+ and HER2- tumor according to American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) or European Society of Medical Oncology (ESMO) guidelines or any national guidelines with criteria conforming to ASCO/CAP or ESMO guidelines.
* Disease progression during or after treatment with an approved cyclin-dependent kinase 4/6 (CDK4/6) inhibitor and endocrine therapy (ET) in the locally advanced or metastatic setting.
* Measurable or non-measurable evaluable, disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Advanced, symptomatic, visceral spread that is at risk of life-threatening complications in the short term appropriate for treatment with cytotoxic chemotherapy at time of entry into the study, as per national or local treatment guidelines.
* Have received more than one-line of therapy for locally advanced or metastatic disease.
* Have received prior chemotherapy for metastatic breast cancer
* Treatment with anti-cancer therapies, including investigational therapies, within 28 days or 5 drug elimination half -lives, whichever is shorter, prior to initiation of study drug. Treatment with an approved oral endocrine therapy (ET) within 7 days prior to initiation of study drug; treatment with fulvestrant or an approved CDK4/6 inhibitor within 21 days prior to initiation of study drug.
* Poor peripheral venous access
* Malabsorption condition or other gastrointestinal (GI) conditions/surgeries that the investigator assesses may significantly interfere with enteral absorption
* History of malignancy within 3 years prior to screening, except for cancer under investigation in this study and malignancies with a negligible risk of metastasis or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence and Severity of Adverse Events (AEs) | Up to 36 months
  Severity of AEs determined according to the CTCAE v5.0 grading scale
Phase Ib: Number of Participants With Dose-Limiting Toxicity (DLTs) | From Day 1 to Day 28 of Cycle 1 (1 cycle=28 days)
Phase II: Progression-free Survival (PFS) | Up to 36 months

SECONDARY OUTCOMES:
Phase Ib: Objective Response Rate (ORR) | Up to 36 months
Phase Ib: Clinical Benefit Rate (CBR) | Up to 36 months
Phase Ib: Area Under the Concentration Time-Curve From Time 0 to Last Measurable Concentration (AUC0-t) of GDC-4198 | Up to 36 months
Phase Ib: Area Under the Concentration Time-Curve From Time 0 to Infinity (AUCinf) of GDC-4198 | Up to 36 months
Phase Ib: Maximum Serum Concentration (Cmax) of GDC-4198 | Up to 36 months
Phase II: ORR | Up to 36 months
Phase II: Duration of Response (DOR) | Up to 36 months
Phase II: CBR | Up to 36 months
Phase II: Overall Survival (OS) | Up to 36 months
Phase II: OS Rate at 6 Months and 12 Months | Month 6, Month 12
Phase II: PFS Rate at 6 Months and 12 Months | Month 6, Month 12
Phase II: Incidence and Severity of Adverse Events (AEs) | Up to 36 months
  Severity of AEs determined according to the CTCAE v5.0 grading scale
Phase II: Plasma Concentration of GDC-4198 | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (8):
  - City of Hope, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center, Irvine, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - City of Hope® Cancer Center Chicago, Zion, Illinois
  - Barbara Ann Karmanos Cancer Institute, Detroit, Maine
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Cancer & Blood Specialists, East Patchogue, New York
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Cancer Research SA, Adelaide, South Australia
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Institut Jean Godinot, Reims, Champagne-Ardenne, France
- Spain (2):
  - Hospital Beata Maria Ana, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing